CLINICAL TRIAL: NCT04003740
Title: Transcranial Direct Current Stimulation for the Treatment of Inattention Symptoms in Attention-deficit/Hyperactivity Disorder: a Randomized, Double-blind, Parallel, Controlled Clinical Trial (TUNED Trial)
Brief Title: TDCS for the Treatment of Inattention Symptoms in Adult ADHD Patients
Acronym: TUNED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-0658
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS (Experimental): The anode will be placed over the right dorsolateral prefrontal cortex (DLPFC) and the cathode over the left DLPFC. Stimulation will be performed for 30 minutes with a current intensity of 2 mA. A ramp-up time of 20 s for the current to go from zero to 2 mA and a ramp-down time that also takes 20 s for the current to go from 2 mA to zero will be used.
  Interventions: Device: Home-based transcranial direct current stimulation
- Sham tDCS (Sham Comparator): The same montage will be used. Sham stimulation will have the same ramp-up and ramp-down time in three different moments (beginning, middle and at the end of the session).
  Interventions: Device: Home-based transcranial direct current stimulation

INTERVENTIONS:
Device: Home-based transcranial direct current stimulation — The stimulation protocol will include one daily stimulation during the first 4 weeks, 2 weekly stimulations for the next 4 weeks, and one weekly stimulation over the last 4 weeks.
  Other Names: Home-based tDCS

SUMMARY:
This study aims at evaluating the efficacy and safety of a home-based tDCS device when compared to a sham stimulation for improving attention in adult ADHD patients.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is a prevalent neurodevelopmental disorder characterized by age inappropriate symptoms of inattention, hyperactivity-impulsivity, or both. The diagnosis of ADHD correlates with several negative outcomes during childhood, adolescence and adulthood, creating huge direct and indirect costs for the health system. The treatment of ADHD involves the use of pharmacologic and non-pharmacologic approaches, and stimulant medications are the most commonly used. Although effective, stimulant medication presents several limitations, reducing long-term adherence. Transcranial direct current stimulation (tDCS) is a neuromodulatory tool that has been shown to be effective for the treatment of various neuropsychiatric disorders. Previous pilot studies applying tDCS in ADHD patients showed conflicting results, and were characterized by heterogeneous methodologies. This study aims at evaluating the effectiveness and safety of tDCS for improving attention in adult ADHD patients by using a more strict methodology, based on a pilot study from our group that showed promising results. Besides that, we aim at exploring the mechanisms of action involved in the effect by using genomic and neuroimaging approaches. By using a computational model, we will also measure the association between clinical response and electric field density propagated with the use of tDCS in brain regions involved in attentional tasks. This will be a phase II-III, parallel, with two intervention groups, randomized, placebo-controlled and double blind study. Only patients without current pharmacological treatment for ADHD will be included in order to evaluate the effectiveness of tDCS as an alternative treatment for the disorder. Patients will be randomized to receive tDCS stimulation with either active or sham home-based devices. The stimulation protocol will include one daily stimulation during the first 4 weeks, 2 weekly stimulations for the next 4 weeks, and one weekly stimulation over the last 4 weeks. After the end of the 12 weeks of stimulation, patients will be followed-up during 6 months in order to observe for how long the effects last. The primary outcome will be obtained after the first 4 weeks of stimulation, with the use of a scale that evaluates inattention symptoms. We hypothesize that the active tDCS will reduce inattention symptoms when compared to sham stimulation, and will result in an increased activation of brain regions related to attention performance. In exploratory analyses, by using genomic approaches, we will observe possible associations between treatment response and specific genes, gene pools and polygenic risk scores. In addition, a functional magnetic resonance imaging test will be performed at rest and during both a sustained attention task (Sustained Attention Test), and a working memory task (N-back Test). This will be performed in order to measure the effects of treatment in the activation of brain regions related to attention performance before and after the first 4 weeks of stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to comply with all requirements of the study;
* Subject is able to provide written consent;
* Subject with an estimated Intelligent Quotient (IQ) score of 80 or above on the Wechsler Adult Intelligence Scale, Third Edition (WAIS-III);
* Subject has a diagnosis of ADHD (combined or inattentive subtypes) according to DSM-V;
* Subject scores 21 points or more in the Clinician Administered ADHD self-report scale - part A (inattention symptoms);
* Subject has not received pharmacological treatment for ADHD during the last month;
* If the subject receives pharmacological treatment for other medical conditions, he/she agrees to maintain the same dosage during the study time;
* Subject is classified as European descendent according to morphologic characteristics, color and ancestry.

Exclusion Criteria:

* Subject has a previous history of neurosurgery;
* Subject has any ferromagnetic metal in the head;
* Subject has implanted medical devices in the head or neck region;
* Subject has a history of non-controlled epilepsy with seizures in the last year;
* Subject has a current depressive episode with a Beck Depression Inventory > 21 points;
* Subject has a current anxiety episode with a Beck Anxiety Inventory > 21 points;
* Subject has a diagnosis of bipolar disorder with maniac or depressive episodes in the last year;
* Subject has a diagnosis of schizophrenia or another psychosis;
* Subject has a diagnosis of autism;
* Subject screened positive for substance use disorder according to The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST);
* Subject has an unstable medical condition with reduction of functional capacity in the next 6 months, like cancer, terminal cardiac disease or terminal pulmonary disease;
* Subject is pregnant or willing to become pregnant in the next 3 months;
* Subject is not able to use a home-based device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Clinician Administered ADHD Self-Report Scale - part A (inattention) at Visit 4 (week 4) | Baseline, Visit 4 (week 4)
  The ADHD Self-Report Scale part A consists of 9 items designed to rate ADHD inattention symptoms. Each item is score from 0 to 4, with a total score ranging from 0 to 36 and higher scores indicating greater symptom severity. The scale will be administered by a clinician with the use of adult prompts.

SECONDARY OUTCOMES:
Clinician Administered ADHD Self-Report Scale - total score | Baseline, Visit 4 (week 4), Visit 5 (week 8), Visit 6 (week 9), Visit 7 (week 10), Visit 8 (week 11), Visit 9 (week 12)
  The ADHD Self-Report Scale consists of 18 items designed to rate ADHD inattention and hyperactivity/impulsivity symptoms. Each item is score from 0 to 4, with a total score ranging from 0 to 72 and higher scores indicating greater symptom severity. The scale will be administered by a clinician with the use of adult prompts.
Behavior Rating Inventory of Executive Functioning - Adult Version (BRIEF-A) | Baseline, Visit 4 (week 4), Visit 5 (week 8), Visit 6 (week 9), Visit 7 (week 10), Visit 8 (week 11), Visit 9 (week 12)
  This is a 75 item self-assessment questionnaire measuring distinct aspects of executive function.
Goal Achievement Scale | Baseline, Visit 4 (week 4), Visit 5 (week 8), Visit 6 (week 9), Visit 7 (week 10), Visit 8 (week 11), Visit 9 (week 12)
  This is a questionnaire created in order to identify specific goals that patients would like to achieve with the proposed intervention, and how much they have achieved from each goal.
N-Back Test | Baseline, Visit 4 (week 4)
  In the N-Back Test subjects are going to be present to a series of letters and required to respond whenever the letter presented is the same as one, two or three before it.
Sustained Attention Test | Baseline, Visit 4 (week 4)
  In the Sustained Attention Tests subjects are required to respond as quickly as possible to a visual stimulus.

OTHER OUTCOMES:
Beck Depression Inventory | Baseline, Visit 4 (week 4), Visit 5 (week 8), Visit 6 (week 9), Visit 7 (week 10), Visit 8 (week 11), Visit 9 (week 12)
  This is a 21 item rating scale for depression symptoms.
Beck Anxiety Inventory | Baseline, Visit 4 (week 4), Visit 5 (week 8), Visit 6 (week 9), Visit 7 (week 10), Visit 8 (week 11), Visit 9 (week 12)
  This is a 21 item rating scale for anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Augusto Rohde, MD-PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schneider M, Ferrazza CP, da Silva Bomber RF, Picon F, Rovaris DL, Sanches PRS, Pereira D, Brunoni AR, Camprodon JA, Caumo W, Bau CHD, Grevet EH, Rohde LA, Leffa DT. Enhancing Goal Achievement in Adults With ADHD: A Participant-Centered Evaluation of Transcranial Direct Current Stimulation From the TUNED Trial. J Atten Disord. 2025 Oct;29(12):1070-1078. doi: 10.1177/10870547251341595. Epub 2025 Jun 17. PMID 40524600
- [Derived] Leffa DT, Grevet EH, Bau CHD, Schneider M, Ferrazza CP, da Silva RF, Miranda MS, Picon F, Teche SP, Sanches P, Pereira D, Rubia K, Brunoni AR, Camprodon JA, Caumo W, Rohde LA. Transcranial Direct Current Stimulation vs Sham for the Treatment of Inattention in Adults With Attention-Deficit/Hyperactivity Disorder: The TUNED Randomized Clinical Trial. JAMA Psychiatry. 2022 Sep 1;79(9):847-856. doi: 10.1001/jamapsychiatry.2022.2055. PMID 35921102